CLINICAL TRIAL: NCT01256710
Title: Trifecta™ Durability Study
Status: Terminated | Type: Observational
Why Stopped: The study was terminated approximately 6 months earlier than planned because 227 subjects (59% more than anticipated) had already completed 10-Year Visits due to lower than expected subject attrition.
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: CS-10-012-EU-TV
Record Dates: First submitted 2010-12-07; First posted 2010-12-08 (Estimated); Results first posted 2023-11-22 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-02

CONDITIONS: Aortic Valve Disease
MeSH Terms: conditions — Aortic Valve Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Trifecta™ Valve Group: Subjects implanted with the Trifecta™ aortic bioprosthesis.
  Interventions: Device: Trifecta™ aortic bioprosthesis

INTERVENTIONS:
Device: Trifecta™ aortic bioprosthesis — Surgical aortic valve replacement with the Trifecta™ valve.

SUMMARY:
The Trifecta™ Durability Study was a multi-center, prospective, single-arm, post-market study conducted in Europe and Canada to collect long-term safety and performance data on the Trifecta™ valve. The Trifecta™ valve is a stented surgical aortic bioprosthesis with bovine pericardial leaflets designed for supra annular placement.

ELIGIBILITY:
Inclusion Criteria:

* Patients implanted for less than 9 months with a Trifecta™ valve, or patients who are candidates for implant with a Trifecta™ valve, as per current guidelines
* Patient requires aortic valve replacement.
* Patient is legal age in host country.
* Patients must be able and willing to provide written informed consent to participate in this investigation
* Patients must be willing and able to comply with all follow-up requirements

Exclusion Criteria:

* Patients with contraindication for cardiac surgery
* Patients who are pregnant.
* Patient is unwilling to or has an inability that reduces his mobility in order to attend the required follow-up visits.
* Patient has active endocarditis
* Patient has had an acute preoperative neurological event defined as patient has not returned to baseline 30 days prior to the planned valve implantation surgery.
* Patient is undergoing renal dialysis.
* Patient has a documented history of substance abuse within one year of enrollment or is currently a prison inmate.
* Patient has a documented thrombus in left atrium or left ventricle.
* Patient had in the past mitral or tricuspid valve replacement.
* Patient needs mitral and/or tricuspid valve replacement.
* Patient has an Ejection Fraction < 25%
* Patient had the Trifecta™ valve implanted as part of this study, but then had the device explanted
* Preoperative evaluation indicates other significant cardiovascular abnormalities such as aortic dissection or ventricular aneurysm.
* Patient has a life expectancy less than two years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients that are candidates for implantation or have been implanted over the past 9 months with a Trifecta™ aortic valve.
Sampling Method: Non-Probability Sample
Enrollment: 1151 (Actual)
Dates: Start 2011-01 (Actual); Primary Completion 2021-03-12 (Actual); Study Completion 2021-03-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sven Lehmann, Principal Investigator — Universitat Herzzentrum Leipzig
Locations (1):
- Universitat Herzzentrum Leipzig, Leipzig, Germany

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Trifecta™ Valve Group
Started | 1151
Completed | 227
Not Completed | 924
Not completed — Death | 449
Not completed — System Explant | 67
Not completed — Transcatheter Aortic Valve-in-Valve Intervention | 28
Not completed — Lost to Follow-up | 67
Not completed — Withdrawal by Subject | 29
Not completed — Physician Decision | 9
Not completed — Subject Noncompliance | 2
Not completed — Study Terminated by Sponsor | 273

BASELINE CHARACTERISTICS:
Population: The analysis population includes participants implanted with the Trifecta™ valve who met all study eligibility criteria and consented to be enrolled in the study.
Arm/Group | Trifecta™ Valve Group
Number analyzed (Participants) | 1151
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.7 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 487
  Male | 664
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Austria | 14
  Belgium | 7
  Canada | 54
  Denmark | 17
  France | 386
  Germany | 404
  Greece | 12
  Italy | 12
  Netherlands | 53
  Norway | 4
  Portugal | 4
  Spain | 153
  Switzerland | 20
  United Kingdom | 11
Baseline Characteristics [Count of Participants; unit: Participants] — NYHA functional classification is a widely used four class ( I, II, III, and IV) measure of the severity of heart failure symptoms. Class I and II patients experience no or slight limitations on their physical activity. Class III and IV patients experience marked limitations on their physical activity or are unable to perform any physical activity without discomfort.
  Participants
    Baseline NYHA III/IV | 566
    History of Coronary Artery Disease | 395
    History of Hypertension | 912
    History of Diabetes | 316
    Previous Cardiovascular Surgery or Procedure | 222
    Concomitant Procedure (e.g., mitral or tricuspid valve repair, CABG, operator reported) | 627
    Concomitant Coronary Artery Bypass Grafting | 360
Implanted Device Size [Count of Participants; unit: Participants]
  19 mm | 115
  21 mm | 335
  23 mm | 411
  25 mm | 222
  27 mm | 57
  29 mm | 11

OUTCOME MEASURES:

1. Primary Outcome: Actuarial Freedom From Reintervention Due to Structural Valve Deterioration
Description: Percentage of participants free from surgical explant or valve-in-valve transcatheter aortic valve intervention for treatment of structural deterioration of the Trifecta™ valve through 10 years post-implant. This percentage is estimated from time-to-event data using the Kaplan-Meier estimator. Structural valve deterioration is deterioration intrinsic to the bioprosthetic valve, due to leaflet calcification, leaflet tears, or other causes, that results in prosthetic valve stenosis or regurgitation.
Time Frame: 10 years
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Trifecta Valve™ Group: Subjects implanted with the Trifecta™ aortic bioprosthesis
Arm/Group | Trifecta Valve™ Group
Number analyzed (Participants) | 1151
percentage of participants | 85.0 [81.6 to 87.8]

2. Secondary Outcome: Actuarial Freedom From All-cause Mortality
Description: Percentage of participants free of death from any cause through 10 years after implant with the Trifecta™ valve, estimated from time-to-event data using the Kaplan-Meier estimator.
Time Frame: 10 years
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Trifecta™ Valve Group
Number analyzed (Participants) | 1151
percentage of participants | 52.2 [48.6 to 55.8]

3. Secondary Outcome: Freedom From Valve Related Mortality
Description: Percentage of participants free from death related to the Trifecta™ valve through 10 years after implant, estimated from time-to-event data using the Kaplan-Meier estimator. Valve-related mortality includes deaths due to any of the following events involving the study valve: structural valvular deterioration, nonstructural valve dysfunction, valve thrombosis, embolism, bleeding events, endocarditis, or reoperation. Sudden, unexplained deaths of participants implanted with the Trifecta™ valve are also counted as valve-related mortality.
Time Frame: 10 years
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Trifecta™ Valve Group
Number analyzed (Participants) | 1151
percentage of participants | 81.6 [78.1 to 84.6]

4. Secondary Outcome: Freedom From Structural Valve Deterioration
Description: Percentage of participants free of structural deterioration of the Trifecta valve through 10 years after implant, estimated from time-to-event data using the Kaplan-Meier estimator. Structural valve deterioration is deterioration intrinsic to the bioprosthetic valve, due to leaflet calcification, leaflet tears, or other causes, that results in prosthetic valve stenosis or regurgitation. The presence of structural valve deterioration is determined by direct visualization of the valve at explant or autopsy or by echocardiographic or other cardiac imaging criteria for assessment of valvular stenosis and regurgitation.
Time Frame: 10 years
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Trifecta™ Valve Group
Number analyzed (Participants) | 1151
percentage of participants | 76.0 [71.9 to 79.6]

ADVERSE EVENTS:
Time Frame: 10 years
Description: Non-serious adverse events had limited analysis during the study focusing on cardiovascular and neurovascular events.
Groups:
- Trifecta Valve Group: Implantation of the Trifecta Valve: Implantation of the bioprothesis valve, Trifecta Valve
Arm/Group | Trifecta Valve Group
All-Cause Mortality (participants affected / at risk) | 449/1151
Serious Adverse Events (participants affected / at risk) | 952/1151
Other Adverse Events (participants affected / at risk) | 562/1151
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Trifecta Valve Group (N=1151)
Blood and Lymphatic System Disorder (Blood and lymphatic system disorders) | 29 (32)
Cardiac disorders (Cardiac disorders) | 533 (937)
Congenital, Familial and Genetic Disorders (Congenital, familial and genetic disorders) | 1 (1)
Ear and Labyrinth Disorders (Ear and labyrinth disorders) | 6 (6)
Endocrine Disorder (Endocrine disorders) | 5 (6)
Eye Disorders (Eye disorders) | 22 (24)
Gastrointestinal Disorder (Gastrointestinal disorders) | 92 (124)
General Disorders (General disorders) | 121 (129)
Hepatobiliary Disorders (Hepatobiliary disorders) | 37 (47)
Immune System Disorders (Immune system disorders) | 1 (1)
Infections and Infestations (Infections and infestations) | 266 (355)
Injury, Poisoning and Procedural Complications (Injury, poisoning and procedural complications) | 101 (114)
Investigations (Investigations) | 4 (4)
Metabolism and Nutrition Disorder (Metabolism and nutrition disorders) | 22 (25)
Musculoskeletal and Connective Tissue Disorders (Musculoskeletal and connective tissue disorders) | 104 (117)
Neoplasms, Benign, Malignant and Unspecified Tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 132 (171)
Nervous System Disorder (Nervous system disorders) | 144 (175)
Product Issues (Product Issues) | 9 (9)
Psychiatric Disorder (Psychiatric disorders) | 35 (39)
Renal and Urinary Disorder (Renal and urinary disorders) | 100 (140)
Reproductive System and Breast Disorder (Reproductive system and breast disorders) | 17 (21)
Respiratory, Thoracic and Mediastinal Disorder (Respiratory, thoracic and mediastinal disorders) | 208 (283)
Skin and Subcutaneous Tissue Disorder (Skin and subcutaneous tissue disorders) | 10 (10)
Social Circumstances (Social circumstances) | 5 (5)
Surgical and Medical Procedures (Surgical and medical procedures) | 21 (22)
Vascular Disorder (Vascular disorders) | 180 (247)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Trifecta Valve Group (N=1151)
Cardiac Disorder (Cardiac disorders) | 389 (518)
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 126 (142)
Vascular disorders (Vascular disorders) | 76 (85)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2010-10-07): https://cdn.clinicaltrials.gov/large-docs/10/NCT01256710/Prot_SAP_000.pdf